CLINICAL TRIAL: NCT00948116
Title: Development of a Biomarker Panel for the Earlier Prediction of Acute Kidney Injury in Patients With Diabetes Mellitus Undergoing Coronary Revascularisation
Brief Title: Development of a Biomarker Panel for the Earlier Prediction of Acute Kidney Injury in Patients With Diabetes
Acronym: BIOMARKERS
Status: Recruiting | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 09/H0703/29; REC 09/H0703/29 (Other: REC); ReDA: 006580 QM (Other: QM)
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus; Renal Impairment
Keywords: Diabetes mellitus; Renal Impairment; Acute Kidney Injury; Coronary revascularisation; eGFR <60ml/min
MeSH Terms: conditions — Diabetes Mellitus; Renal Insufficiency; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine samples will be retained for the duration of the study
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Diabetes mellitus, renal impairment: Patients with both diabetes mellitus and eGFR <60 ml/min

SUMMARY:
Patients living with diabetes mellitus have double the risk of kidney failure compared to patients without diabetes following use of dye in many x-rays and procedures to diagnose and treat narrowing of the arteries (blood vessels) in the heart that can lead to angina or a heart attack. Heart disease is the commonest cause of death in patients with diabetes. People with diabetes are more likely to need these tests/treatments. By identifying those at greater risk of kidney complications we may be able to make these tests/treatments safer and offer them to more patients with diabetes.

DETAILED DESCRIPTION:
Diabetes mellitus is an important risk factor for the development of contrast induced nephropathy (CIN), acting as a 'risk multiplier', amplifying the risk of acute kidney injury in these patients. There are important prognostic implications following the development of CIN and it is associated with a significantly increased mortality at 1 year. Diabetes is a major risk factor for coronary disease and these patients often have significant co-morbidities.

Currently creatinine is used to assess risk but this often lags behind clinical status. There is a pressing need for the development of novel, specific biomarkers to improve the detection and treatment of CIN and improve patient outcome in this high risk population.

This is a single centre,study in diabetic patients already undergoing a planned procedure, that is, a percutaneous coronary intervention (PCI). They are patients who are deemed to have an enhanced risk of contrast induced nephropathy by virtue of their diabetic and renal status, the latter being defined by a reduced eGFR which is a marker of renal disease and is based on the creatinine and characteristics of the patient. No additional interventions that are not part of their routine clinical care will be undertaken in these patients. We will be identifying natural biomarkers by obtaining serum and urine samples from these patients.

From a retrospective audit of the cardiac catheter lab database and a review of the literature we have estimated that a sample size of approximately 250 patients with DM and CKD (eGFR < 60 ml/ml) will be needed. We envisage that that we will encounter at least 50 cases of CIN from this cohort. (based on an expected incidence of CIN between 15-30% in this group). Looking for a study rate difference of at least 25%, for power of 95% and confidence intervals of 95% (with Fleiss correction) we will need at least 204 evaluable patients (to avoid Type 2 error). In view of potential drop-out of 10-15% we therefore intend to recruit 250 patients By using C statistics (Receiver operator curve analysis) we will be able to confirm or otherwise that either a particular biomarker or a combination of several biomarkers within 18 hours of procedure will increase the predictive power of CIN developing 72 hours later.

As part of their normal care patients will arrive in hospital on the morning of their planned PCI. They will at some point during the day undergo their PCI. Blood and urine will be taken just prior to the procedure and then at 2 hours, 4 hours, 8 to 12 hours, pre discharge and 3 days after the PCI.

We will then analyse the samples using ELISA techniques and correlate the biomarkers with creatinine to explore which biomarkers or panel of biomarkers may be able to diagnose contrast induced nephropathy earlier than creatinine can currently.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years, known diabetes mellitus or BM on arrival consistent with probable diagnosis of diabetes, eGFR <60 ml/min
2. Undergoing a PCI procedure
3. Agrees to the additional collection of blood and urine samples as outlined above
4. Agrees to access of their clinical records for the collection of relevant medical data
5. No history or signs of drug abuse
6. Able to understand and sign the written Informed Consent Form
7. Able and willing to follow the Protocol requirements

Exclusion Criteria:

1. Cardiogenic shock
2. Pregnancy
3. Patient on renal replacement therapy (haemodialysis/CAPD/renal transplant)
4. Known clinically significant infection such as HIV, Hepatitis or TB
5. Any patient determined not able to make a reasoned, informed consent prior to the planned interventional procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetes mellitus and renal impairment
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2009-06-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Development of contrast induced nephropathy (CIN) which will be defined as an increase in Cr of ≥ 44 μmol/l within 72 hours post-procedure. | up to 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: AKHIL KAPUR, Principal Investigator — CONSULTANT CARDIOLOGIST AND HONORARY SENIOR LECTURER, BARTS AND THE LONDON NHS TRUST; KATIE QURESHI, Principal Investigator — Clinical Research Fellow/Specialist Registrar, Barts and The London NHS Trust; MAGDI YAQOOB, Principal Investigator — PROFESSOR AND CONSULTANT NEPHROLOGIST, HEAD DEPARTMENT OF EXPERIMENTAL MEDICINE AND NEPHROLOGY
Locations (1):
- The London Chest Hospital, London, United Kingdom